CLINICAL TRIAL: NCT06266442
Title: Longitudinal Assessment of Clinical Pulmonary Mycobacterium Avium Isolates in Treated Patients Using Whole Genome Sequencing
Brief Title: M. Avium WGS During Mav-PD Treatment
Status: Recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Western University, Canada (Other); Public Health Ontario Laboratory, Canada (Unknown)
Responsible Party: Principal Investigator, Theodore (Ted) Marras, Director, Toronto Western Hospital / University Health Network Nontuberculous Mycobacterial Disease Program, Principal Investigator, Associate Professor, University Health Network, Toronto
Other Study IDs: Mav-WGS
Record Dates: First submitted 2023-12-27; First posted 2024-02-20 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Mycobacterium Avium; Mycobacterium Infections, Nontuberculous; Mycobacterium Infections; Nontuberculous Mycobacterial Lung Disease; Respiratory Tract Diseases
Keywords: Nontuberculous mycobacterium; Whole genome sequencing; Mycobacterium avium
MeSH Terms: conditions — Mycobacterium avium-intracellulare Infection; Mycobacterium Infections, Nontuberculous; Mycobacterium Infections; Respiratory Tract Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sputum and environmental samples, DNA extracts from NTM derived from the patients and their environments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Whole genome sequencing testing — Whole genome sequencing

SUMMARY:
This is a prospective observational study using whole genome sequencing (WGS) to investigate whether new strains (other than the initially identified strain(s)) of M. avium are responsible for persistently culture positive sputum during treatment (refractory disease), or the reversion to culture positive sputum after prior conversion to negative. The study will further investigate for differences between participants living in the Toronto/York region versus participants living elsewhere.

The primary goal of this prospective observational study is to understand why some patients with M. avium lung disease have persistent or recurrent M. avium in their sputum despite treatment. The aim is to understand whether it is usually due to treatment failure or new infection.

DETAILED DESCRIPTION:
Mycobacterium Avium complex (MAC) are a subset of nontuberculous mycobacteria (NTM) that are typically found in the soil and water and can cause pulmonary lung disease. Treatment of MAC is challenging as it typically requires the use of three or more antibiotics for over a long period of time and the rate of eradication is suboptimal.

Mac-WGS is an observational study that aims to understand whether new strains of M. avium are responsible for persistently culture-positive sputum during treatment. Whole genome sequencing (WGS) will be performed on M. avium isolates from the sputum of patients with Mav-PD, over the duration of the study. Additionally, home environmental samples will be collected and sequenced to identify any home source of infection.

As an observational study, participants will receive routine standard of care treatment as per discretion of the physician. Standard of care includes monthly sputum submissions. The M. avium isolated from the sputum before treatment and every three months while on treatment (until such time that the sputum becomes culture-negative) will be analyzed by WGS. If sputum becomes culture-positive again, the isolated germ will also be analyzed by whole genome sequencing. It will be determined whether the identical strain of M. avium is always present or whether more than one strain is present which would suggest either multi-strain infection or the acquisition of new strains of M. avium while on treatment. Additionally, participant's home environmental samples (i.e. faucets and showerhead biofilms) will be cultured to determine whether M. avium can be recovered and if so, it will be analyzed with WGS to assess whether it is the same strain as in the participant's sputum.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Willing to provide informed consent and participate in study procedures
* Residing continuously in Ontario during the past five years
* Mav-PD, either initial or recurrent (previously treated patients will be eligible) five years
* Meet American Thoracic Society (ATS) / Infectious Diseases Society of America (IDSA) NTM disease criteria for Mav-PD

Exclusion Criteria:

* Lack of an available pre-treatment M. avium isolate in the PHOL isolate bank
* The inability to produce sputum either spontaneously or by induction with nebulized hypertonic saline
* Cavitation >3 cm internal diameter
* Known macrolide-resistant MAC infection
* HIV infection
* Known diagnosis of cystic fibrosis
* History of solid organ or hematological transplantation
* Severe comorbid illness that is reasonably expected to limit survival to <24 months
* Residing in mid/north York region (King, Aurora, Newmarket, Whitechurch-Stouffville, East Gwillimbury or Georgina)
* Having moved between regions (Toronto/southern York region vs non-Toronto/York region vs mid-northern York region) within the past 5 years

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients at the Toronto Western Hospital (TWH) Nontuberculous Mycobacterial (NTM) clinic who are to be initiated on therapy for Mav-PD.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-05-13 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with persistent culture-positive sputum despite antimicrobial therapy | 24 months
  Whole genome sequencing

SECONDARY OUTCOMES:
Whether patients with Mav-PD have evidence of polyclonal infection as demonstrated by the presence of >1 strain of M. avium in the pre-treatment sputum or a sputum sample during treatment | 24 months
  Whole genome sequencing
Whether there is a source of infection from the home water environment | 24 months
  M. avium strains from sputum and home water source samples will determined through WGS analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Marras, MD, Principal Investigator — UHN
Locations (1):
- University Health Network, Toronto, Ontario, Canada